CLINICAL TRIAL: NCT02843217
Title: Innovations in Enhancing Colorectal Cancer Screening
Brief Title: Regional Native American Community Networks Program (RNACNP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Dedra Buchwald, Human Subjects Protection Manager, Washington State University
Model: Crossover | Purpose: Screening
Other Study IDs: U54CA153498 (NIH)
Record Dates: First submitted 2016-06-15; First posted 2016-07-25 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2016-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text Messaging (Experimental)
  Interventions: Behavioral: Lifestyle, screening

INTERVENTIONS:
Behavioral: Lifestyle, screening

SUMMARY:
Aim: Determine the overall effectiveness of a targeted digital messaging intervention at improving colorectal cancer (CRC) screening rates compared to care as usual.

Hypothesis: Screening rates will be higher for patients who receive the digital messaging intervention, compared to the control group in which patients receive care as usual.

DETAILED DESCRIPTION:
Native People for Cancer Control is one of the projects under Partnerships for Native Health, and is 1 of 23 Community Networks Programs funded by the National Cancer Institute. The aim of Native People for Cancer Control is to reduce cancer health disparities by conducting training, research, education and outreach, in collaboration with American Indian and Alaska Native communities. We do this work in partnership with Native people, communities, and organizations in an 8-state area, including: Alaska, Washington, Wyoming, Oregon, Idaho, Montana, North Dakota, and South Dakota. Our program consists of 4 cores:

Administrative Core: assists with grant administration, budgeting, sub-contracts with Tribes, program planning, and reporting.

Outreach/Education Core: assists with cancer education, outreach, health promotion, and cancer prevention activities among urban and rural AI/AN people.

Training Core: builds capacity for Native faculty-level investigators, and students, to conduct research.

Research Core: conducts community-based participatory research on colorectal cancer screening, health literacy, health communication, and cancer risk factors among American Indian and Alaska Native people.

The main research project under Native People for Cancer Control is titled, "Innovations in Enhancing Colorectal Cancer Screening". The goal of this project is to develop, implement, and evaluate a community wide, multi-media campaign to improve colorectal cancer screening among American Indians and Alaska Natives in 3 communities.

ELIGIBILITY:
Inclusion Criteria:

* AI/AN
* Age 50-75
* Active clinical patient

Exclusion Criteria:

* Not AI/AN

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2010-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening, beginning age 50 | 9 month intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Pullman, Washington, United States